CLINICAL TRIAL: NCT03186469
Title: Generations in Families Talking Safe Sleep
Acronym: GIFTSS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Arkansas Children's Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: 203247
Record Dates: First submitted 2017-06-12; First posted 2017-06-14 (Actual); Last update posted 2019-07-18 (Actual); Status verified 2019-07

CONDITIONS: Sudden Infant Death
MeSH Terms: conditions — Sudden Infant Death | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Data collector will be blinded as to which arm study participants are enrolled
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Behavioral: Safety Baby shower Teen Only (Active Comparator): Only the teen will receive the educational intervention.
  Interventions: Behavioral: Safety Baby shower
- Behavioral: Safety Baby shower Dyad (Active Comparator): Both the teen and the teens support person will receive the educational intervention.
  Interventions: Behavioral: Safety Baby shower
- Behavioral: Standard of Care Control (Other): Standard of care.
  Interventions: Behavioral: Standard of Care

INTERVENTIONS:
Behavioral: Safety Baby shower — A Safety Baby Shower using didactic and experiential teaching methods to educate participants on safety topics focused on reducing infant mortality. Participants receive safety products as their "shower gifts" with education on appropriate use of the products. The relaxed setting also encourages participants to seek answers and clarify myths from credible sources not otherwise available among family and friends. For intervention provides information on the infant's sleep position, bedding, co-sleeping, and tobacco exposure, all of which, alone or in combination, are risk factors for sleep-related deaths in infants. Breastfeeding, a protective factor for SIDS, will be encouraged.
  Arms: Behavioral: Safety Baby shower Dyad; Behavioral: Safety Baby shower Teen Only
Behavioral: Standard of Care — Participants will received standard of care in regards to infant injury prevention. Written material on car seat safety, prevention of abusive head trauma, and safe sleep environments will be provide to participants.
  Arms: Behavioral: Standard of Care Control

SUMMARY:
Teen mothers present a unique set of challenges in reducing the risk for sleep-related infant mortality, in part because they may not be the sole decision-maker for an infant's sleep environment and position and they make seek advice from older female support people. Investigators will conduct a randomized controlled trial of a educational intervention to mitigate the risks of unsafe infant sleep practices across generations. Given the complexity and variability of teen-SCG relationships, investigators will include an examination of inter- and intra-personal factors that are key control variables or may mediate the uptake of safe sleep recommendations. Investigators believe that the intervention will empower support people to positively influence a teen mother's adoption of safe sleep recommendations.

DETAILED DESCRIPTION:
The infant mortality rate in the United States (US) is 6.14 per 1000-a rate higher than most other developed countries. Sudden Infant Death Syndrome (SIDS) and suffocation account for more than half of all Sudden Unexpected Infant Deaths (SUID) and represent the first and third leading causes of post neonatal infant death (death in an infant age 28 days to 1 year) in the US. The importance of SIDS and SUID is reflected by strategic planning efforts conducted by the NICHD over the past two decades. Young, poor, unmarried, and minority women are at elevated risk for SIDS. Infants born to mothers aged 15 - 19 are at increased risk for infant mortality in general, with a rate of 9.59 per 1000 in 2008. National surveys including the National Infant Sleep Position Study and the Pregnancy Risk Assessment Monitoring System show that teen mothers are less likely to adhere to recommendations for supine sleeping, bed surfacing (including bed sharing on an adult bed) and other environmental precautions. Teen mothers present a unique set of challenges in reducing the risk for sleep-related infant mortality, in part because they may not be the sole decision-maker for an infant's sleep environment and position. Teens often rely on their own mother or other senior caregivers (SCG) for information and assistance with child care. For the proposed study, SCG influence on a key set of parenting behaviors is especially salient. Several studies have demonstrated the important role of SCG on maternal behavior related to infant safety, breastfeeding, and sleep environment and practices. Attitudes about sleep position have been found to be more strongly associated with appropriate behaviors than knowledge. A mother's beliefs about choking risks have been found to be significant determinants of supine sleep positions, but those beliefs can be influenced by the source and dosage of advice. The infant's grandmother or other SCG can influence a mother's decision on sleep position. Other evidence indicates that the SCG to whom a teen mother may turn to for advice may also fail to adhere to recommendations for safe sleep. For this study investigators propose to build upon an existing, well-received Safety Baby Showers (SBS) educational program. The standardized intervention (which is currently utilized in 10 counties in Arkansas to educate pregnant mothers) uses engaging activities to educate participants on infant safety topics focused on motor vehicle safety, home safety, and safe sleep. The Central Hypotheses are as follows: H1) Teen mothers exposed to an intensive educational intervention will be more likely than controls to appropriately adopt safe sleep practices (supine position and in an appropriate sleep environment) with their infants, and H2) Because teen mothers will model their choice of infant sleep position and environment on behavior of their mothers or other significant female senior caregivers, they will be more likely to use those safe sleep practices when they and their mothers or other significant female senior caregivers also participate in tailored education about safe infant sleep. In order to accomplish the NIH funded research project investigators will proceed with three phases. Phase 1: Preparatory- Investigators will further refine the existing infant sleep safety intervention for pregnant teens and their mothers or other identified significant female SCGs and Phase 2: Pilot-Investigators will pilot the refined infant sleep intervention, recruitment strategies, and data collection methods and refine as needed based on pilot participant feedback. Phase 3: Full Launch- Investigators will conduct a randomized controlled trial to determine if the educational intervention both with and without SCGs is associated with an increase in both knowledge of appropriate safe sleep behaviors and in observed supine infant sleep positioning and appropriate sleep environment among teen mothers. Full Launch- Investigators will conduct a randomized controlled trial to determine if the educational intervention both with and without SCGs is associated with an increase in both knowledge of appropriate safe sleep behaviors and in observed supine infant sleep positioning and appropriate sleep environment among teen mothers

ELIGIBILITY:
Inclusion Criteria:

* First child
* Live in Faulkner, Saline, White, Pulaski, Jefferson, Lonoke County
* 13-28 weeks pregnant
* Teen identified female support person age 30 or older

Exclusion Criteria:

* Non English speaking
* No support person identifiable

Ages: 13 Years to 19 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 146 (Actual)
Dates: Start 2014-10-07 (Actual); Primary Completion 2020-04-30 (Estimated); Study Completion 2020-10-31 (Estimated)

PRIMARY OUTCOMES:
Use of safe sleep environment | 2-3 months post delivery
  comparison of safe vs unsafe sleep

CONTACTS AND LOCATIONS:
Overall Officials: Mary E Aitken, MD, MPH, Principal Investigator — Arkansas Children's Hospital Research Institute
Locations (1):
- Arkansas Children's Research institute, Little Rock, Arkansas, United States

IPD SHARING:
Plan to Share IPD: No